CLINICAL TRIAL: NCT02921529
Title: Perioperative Transcutaneous Electrical Acupoint Stimulation for Enhanced Recovery After Laparoscopic Colon Surgery:a Multi-center Randomized Controlled Clinical Trial
Brief Title: TEAS Enhanced Recovery After Laparoscopic Colon Surgery
Acronym: ARCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Doctor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-2016-09-01
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Recovery
Keywords: Postoperative recovery; colon surgery
MeSH Terms: interventions — Acupuncture Therapy; Electric Stimulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Inventions were given by an investigator who is not involved in patient care. The anesthetists, surgeons,staff in the ward, the one who record the outcomes, and data analyzer were all blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEAS (Experimental): Patients were given 30min of TEAS(transcutaneous electrical acupoint stimulation) before anesthesia and 1,2,3 day after surgery
  Interventions: Other: TEAS
- false stimulation (Sham Comparator): Attach electrodes without electric current
  Interventions: Other: false stimulation

INTERVENTIONS:
Other: TEAS — Electric stimulation was given through electrode attached to specific acupoints
  Other Names: Acupuncture; Electric stimulation
  Arms: TEAS
Other: false stimulation — Electrodes were attached to specific acupoints without electric current
  Other Names: sham stimulation
  Arms: false stimulation

SUMMARY:
The purpose of this study is to observe the effects of transcutaneous electrical acupoint stimulation(TEAS) on postoperative recovery after laparoscopic colon surgery.

DETAILED DESCRIPTION:
Patients were randomly assigned to two groups, receiving TEAS andno stimulation respectively. Interventions were given 30min before anesthesia and 1, 2 , 3 day after surgery, lasted 30min each time . The acupoints of TEAS group are bilateral ST36/SP6 combined with PC6/LI4, and the control group only attach electrodes without electric current. The frequency of TEAS is set to 2/10 Hz. After surgery, the time of meeting discharge criteria, first flatus and defecation were recorded. Score of PONV, life quality, sleep quality and VAS of pain were evaluated 24, 48 and 72h after surgery. The postoperative complications, re-exploration, cost of hospitalization and adverse events were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 75 years old；
* ASA I-III；
* Scheduled for elective laparoscopic colon surgery under general anesthesia；
* BMI between 18 and 30；
* Informed consented.

Exclusion Criteria:

* Patients with contraindications to the use of electroacupuncture, such as skin damage or infection at the acupoints；
* Patients with difficulty in communication；
* Emergency surgery；
* Patients who are with distant metastasis;
* Patients who are with history of myocardial infarction or cerebral infarction in the past six months；
* Patients who are with long history of taking NSAIDS，hormone or immunosuppressive agents；
* Patients who are recruited in other clinical trials in the last 3 months；
* Other situations researcher think shouldn't be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Time to meeting discharge criteria | end of the surgery to discharge,with an average of 7 days

SECONDARY OUTCOMES:
Time to first flatus | end of the surgery to discharge,with an average of 7 days
Time to first defecation | end of the surgery to discharge,with an average of 7 days
Incidence of postoperative complications | end of the surgery to discharge,with an average of 7 days
Time to first oral intake of water | end of the surgery to discharge,with an average of 7 days
visual analogue scale | end of surgery to 24 hours, 48 hours, and 72 hours after surgery
  0 is for no pain, 10 is for pain that can not be tolerated
incidence of nausea and vomiting | end of surgery to 24 hours, 48 hours, and 72 hours after surgery
quality of sleeping score | end of surgery to 24 hours, 48 hours, and 72 hours after surgery
  0 is for totally insomnia, 10 is for perfect sleep
quality of recovery | end of surgery to 24 hours, 48 hours, and 72 hours after surgery
  using a questionaire including 15 items that covering postoperative recovery
expense | end of the surgery to discharge,with an average of 7 days
  patients' cost after surgery

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - First Afiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Tongji Hospital, Wuhan, Hubei
  - Xijing Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR